CLINICAL TRIAL: NCT02994537
Title: Study of the Clinical Features of Autoimmune Hepatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li Yang (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Li Yang, MD, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: AAIH-001
Record Dates: First submitted 2016-12-02; First posted 2016-12-16 (Estimated); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Hepatitis, Autoimmune
Keywords: autoimmune hepatitis, diagnosis, pathogenesis, treatment, prognosis
MeSH Terms: conditions — Hepatitis, Autoimmune; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and or liver tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- acute autoimmune hepatitis: Patients diagnosed autoimmune hepatitis(AIH) are divided into acute cohort or chronic cohort (acute-on-chronic and chronic were all included)by biochemical results, such as liver function and coagulation, then the investigators will compare the histological results, treatment effects and prognosis between the two groups. Further more, the investigators will study the pathogenesis of different forms of autoimmune hepatitis. Even more, the investigators want to explore drug induced AIH and viral hepatitis related AIH.
  Interventions: Other: Different biochemical results or pathogenesis.

INTERVENTIONS:
Other: Different biochemical results or pathogenesis. — Comparing the pathogenesis,clinical characteristics and treatment effects between the acute autoimmune hepatitis group and the chronic autoimmune hepatitis group. The investigators don't use special intervention.

SUMMARY:
The purpose of this study is to explore the pathogenes, clinical characteristics, laboratory and histological examination results, treatment and prognosis of autoimmune hepatitis(AIH). At phase 1, the investigators focus on studying of the clinical characteristics of acute autoimmune hepatitis, and then will study the difference about treatment effects between acute autoimmune hepatitis and chronic AIH. Morever, the investigators have noticed that drug induced AIH have some special characteristics that may be beneficial to distinguish it with durg induced liver disease. Therefore the investigators will do some studies about drug induced AIH or other disease which maybe related to the onset of AIH.

DETAILED DESCRIPTION:
Now this study has been researched at phase 1, the investigators focus on studying the difference between acute AIH and chronic AIH. In this phase, the investigators analysed the serum biochemical results such as ALT,AST,IgG,PT,INR and so on, and also compared the histological performance. Finally, we compared the percentages of biochemical remission in the two groups, and the time from initial treatment to biochemical remission has also been put into the analysis. Now, the investigators are preparing for submitting the manuscript of phase 1.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of autoimmune hepatitis

Exclusion Criteria:

* Other causes of liver disease, such as viral hepatitis, drug induced liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, overlap syndrome and so on.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from the hospital outpatient or inpatient department, there is no geographical restrictions.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical remission of participants | 3 years after standard immunosuppressive treatment.
  This study is now in the phase 1, and the outcome at phase 1 is the biochemical remission of AIH patients. In details, if the participants' serum ALT,AST and IgG returned to normal, that means this participant reached the biochemical remission.

CONTACTS AND LOCATIONS:
Overall Officials: Li Yang, MD, Study Director — Division of Gastroenterology & Hepatology,West China Hospital,Sichuan University
Locations (1):
- Division of Gastroenterology & Hepatology,West China Hospital,Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
The investigators need to discuss with other participants whether or not to share data of the study.

REFERENCES:
- [Background] Kessler WR, Cummings OW, Eckert G, Chalasani N, Lumeng L, Kwo PY. Fulminant hepatic failure as the initial presentation of acute autoimmune hepatitis. Clin Gastroenterol Hepatol. 2004 Jul;2(7):625-31. doi: 10.1016/s1542-3565(04)00246-0. PMID 15224287
- [Result] Fujiwara K, Nakano M, Yasui S, Okitsu K, Yonemitsu Y, Yokosuka O. Advanced histology and impaired liver regeneration are associated with disease severity in acute-onset autoimmune hepatitis. Histopathology. 2011 Apr;58(5):693-704. doi: 10.1111/j.1365-2559.2011.03790.x. Epub 2011 Mar 14. PMID 21401703
- [Result] Abe M, Hiasa Y, Masumoto T, Kumagi T, Akbar SM, Ninomiya T, Matsui H, Michitaka K, Horiike N, Onji M. Clinical characteristics of autoimmune hepatitis with histological features of acute hepatitis. Hepatol Res. 2001 Nov;21(3):213-219. doi: 10.1016/s1386-6346(01)00109-7. PMID 11673106
- [Derived] Shen Y, Lu C, Men R, Liu J, Ye T, Yang L. Clinical and Pathological Characteristics of Autoimmune Hepatitis with Acute Presentation. Can J Gastroenterol Hepatol. 2018 Mar 18;2018:3513206. doi: 10.1155/2018/3513206. eCollection 2018. PMID 29744332